CLINICAL TRIAL: NCT01182311
Title: Duration of Long-Term Immunity After Hepatitis B Virus Immunization
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100187; 10-DK-0187
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Virus; Hepatitis B Vaccine; Immunity; B-Cell Response; T-Cell Response; Hepatitis B Immunity; Hepatitis B Virus Vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (6):
- Controls: Never received HBV vaccine and never had HBV
- HIV vaccinated >= 10 years: Well compensated HIV disease, vaccinated HBV >= 10 years ago
- Spontaneously recovered >= 10 years: Spintaneously recovered from acute HBV >= 10 years ago
- Vaccinated >= 20 years: Vaccinated against HBV >= 20 years ago
- Vaccinated 10 < 15 years: Vaccinated against HBV 10 < 15 years ago
- Vaccinated 15 < 20 years: Vaccinated against HBV 15 < 20 years ago

SUMMARY:
Background:

* The hepatitis B vaccine has been shown to be safe and effective in preventing transmission of the hepatitis B virus. Response rates to the initial three doses of the vaccine are high, with significant or even complete immune response. However, this level has been reported to decline rapidly within the first year and more slowly thereafter. There is little data on the durability and long-term protection provided by the hepatitis B vaccine administered to adults in the United States.
* Vaccinated individuals are believed to be protected against hepatitis B virus infection because of a memory immune response. Even if antibody levels are low, the immune system will still be able to produce enough antibody to neutralize the hepatitis B virus. Therefore, booster doses of the vaccine are not recommended, except for some high-risk individuals such as patients on dialysis. Researchers are interested in determining the durability of the immune response of the hepatitis B vaccine in adults with low or intermediate risk for hepatitis B virus infection.

Objectives:

- To examine the long-term immune status of human immunodeficiency virus (HIV) positive and negative individuals who received the hepatitis B vaccine during adulthood, compared with the immune status of individuals who acquired natural immunity by recovering from acute hepatitis B during adulthood.

Eligibility:

* Individuals at least 18 years of age who were vaccinated against hepatitis B at least 10 years ago.
* Individuals at least 18 years of age who contracted and recovered from acute hepatitis B at least 10 years ago.
* Individuals at least 18 years of age who have well-controlled HIV and were vaccinated against hepatitis B at least 10 years ago.

Design:

* Participants will have a single outpatient study visit and potential follow-up visits as part of this protocol.
* Participants will complete a questionnaire assessing possible risk factors for hepatitis B infection, and will provide blood samples to test for hepatitis B antibodies and other immune system studies.
* Participants will receive a letter or phone call with the results of the blood tests:
* Those who no longer have protective levels of antibody against the hepatitis B virus will be offered a booster dose of the hepatitis B vaccine. To monitor immune response to the booster vaccine, additional study visits will be scheduled at 1 and 3 weeks following the booster.
* Those who have chronic infection with the hepatitis B virus will be advised to follow up with their primary care physician, and may be eligible to participate in ongoing treatment trials for chronic hepatitis B.
* Those who have abnormal blood tests will be referred back to their primary care physician for investigation of the abnormal tests results, and may also be referred to other National Institutes of Health protocols.
* Additional tests will evaluate immune response to the measles, mumps, and rubella (German measles) viruses. Some participants may be advised to have an additional MMR vaccine through their primary care physician.

DETAILED DESCRIPTION:
Hepatitis B vaccine is very effective at preventing infection with the hepatitis B virus (HBV). Several studies have reported on the long-term efficacy of the HBV vaccine and indicate a decline in titers of antibody against hepatitis B surface antigen (anti-HBs) over time. However, most of these studies were performed in persons vaccinated as infants or children. This protocol is designed to examine the long-term immune status of HIV positive and negative individuals who were vaccinated during adulthood, and to compare it to the immune status of individuals who acquired natural immunity by recovering from acute hepatitis B during adulthood. Individuals who lost the vaccine-induced humoral immune response, will be offered a booster vaccination and their immune response to the booster vaccination will be assessed. In this study, we will recruit 150 subjects who were vaccinated secondary to their job-related risk of acquiring HBV infection. An additional 50 subjects who had spontaneously recovered from acute hepatitis B (Bullet) 10 years ago, 50 patients with well-compensated HIV infection who received HBV vaccine (Bullet) 10 years ago and 10 subjects who were never vaccinated and never infected with the hepatitis B virus will be enrolled as comparison groups. All subjects will be asked to complete a questionnaire to assess their HBV exposure risk as well as factors that may affect their immune response. Immunological assays include the quantitation of HBV-specific antibodies and the qualitative and quantitative assessment of HBV-specific memory B cells and T cells at the indicated time intervals after vaccination or after recovery from acute hepatitis B. Additional immunological assays include testing for antibody to measles, mumps and rubella (German measles) viruses to compare the longevity of antibody response to these vaccines or natural infection to the antibody response to the hepatitis B vaccine or natural infection. The results of this study will help to answer the question whether a booster vaccination is required and at which time after the primary vaccination course it should be considered.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years or above and < 60 years when the first dose of hepatitis B vaccine was administered
  2. Male or female
  3. Vaccination with 3 doses of either plasma-derived or recombinant HBV vaccine within one year (with the exception of the 10 patients who were never vaccinated and never infected with the hepatitis B virus)
  4. Vaccinated subjects must be able to provide written documentation indicating the dates of their hepatitis B immunization series. In the absence of written documentation, subjects will be asked to sign a written affidavit obtained either from themselves or their physician stating the date of vaccination accurate to one year and that they did not receive a booster dose to the best of their knowledge.
  5. For recovered patients, spontaneous recovery from acute hepatitis B must have occurred prior to the year 2000
  6. Willing and able to provide written, informed consent

Additional Inclusion Criteria for HIV positive cohort

1. CD4 count of great than or equal to 250 /mm3 at time of vaccination
2. Known HIV infection at time of vaccination

EXCLUSION CRITERIA:

1. History of chronic HBV infection
2. Incomplete HBV vaccine doses (with the exception of the 10 patients who were never vaccinated and never infected with the hepatitis B virus)
3. Known non-response to an adequate course of hepatitis B vaccine
4. Received a booster dose of HBV vaccine
5. Current or recent (within the last 1 year) use of immunosuppressive/immuno-modifying agents
6. Use of immunosuppressive/immuno-modifying agents at the time of vaccination
7. Renal failure with requirement for dialysis
8. Anti-HIV positive (Except for HIV positive cohort)
9. Anti-HCV positive
10. History of bone marrow or stem cell transplant
11. History of organ transplant
12. Known underlying immune suppressive condition
13. Subjects with clinically significant anemia, hemoglobin <10g/dL will be excluded from participating in the assessment of response to a booster dose of HBV vaccine until their hemoglobin is greater than or equal to12g/dL.
14. Anti-HBc positivity for the 10 patients who were never vaccinated and never infected with the hepatitis B virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital employees
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Protective Anti-HBs | At start of study
  Anti-HBs levels >12 mIU/mL

SECONDARY OUTCOMES:
HBV-specific antibodies | At start of study
Quantitative assessment of HBV-specific memory B cells and T | At start of study

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dienstag JL. Hepatitis B virus infection. N Engl J Med. 2008 Oct 2;359(14):1486-500. doi: 10.1056/NEJMra0801644. No abstract available. PMID 18832247
- [Background] Kim WR. Epidemiology of hepatitis B in the United States. Hepatology. 2009 May;49(5 Suppl):S28-34. doi: 10.1002/hep.22975. PMID 19399791
- [Background] McQuillan GM, Coleman PJ, Kruszon-Moran D, Moyer LA, Lambert SB, Margolis HS. Prevalence of hepatitis B virus infection in the United States: the National Health and Nutrition Examination Surveys, 1976 through 1994. Am J Public Health. 1999 Jan;89(1):14-8. doi: 10.2105/ajph.89.1.14. PMID 9987458
- [Derived] Gara N, Abdalla A, Rivera E, Zhao X, Werner JM, Liang TJ, Hoofnagle JH, Rehermann B, Ghany MG. Durability of antibody response against hepatitis B virus in healthcare workers vaccinated as adults. Clin Infect Dis. 2015 Feb 15;60(4):505-13. doi: 10.1093/cid/ciu867. Epub 2014 Nov 10. PMID 25389254
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-DK-0187.html